CLINICAL TRIAL: NCT03821480
Title: AN OPEN-LABEL, RANDOMIZED, SINGLE DOSE, CROSSOVER PIVOTAL BIOEQUIVALENCE STUDY OF FLUCONAZOLE CAPSULE 50 MG IN HEALTHY ADULT SUBJECTS
Brief Title: Diflucan Bioequivalence Study For Transferring The Manufacture
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A0561026
Record Dates: First submitted 2019-01-28; First posted 2019-01-29 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Bioequivalence
Keywords: Fluconazole
MeSH Terms: interventions — Drug Evaluation; Fluconazole

STUDY DESIGN:
Intervention Model Description: open-label, randomized, single dose, 2-treatment, 2-period crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluconazole 50 mg, Manufacturer: Amboise (Experimental): Test drug
  Interventions: Drug: Test drug
- Fluconazole 50mg, Manufacturer:West Ryde (Active Comparator): Reference drug
  Interventions: Drug: Reference drug

INTERVENTIONS:
Drug: Test drug — Fluconazole capsule 50 mg Manufacturer: West Ryde
  Other Names: Fluconazole capsule 50mg
  Arms: Fluconazole 50 mg, Manufacturer: Amboise
Drug: Reference drug — Fluconazole capsule 50 mg Manufacturer: Amboise
  Other Names: Fluconazole capsule 50mg
  Arms: Fluconazole 50mg, Manufacturer:West Ryde

SUMMARY:
This study is to assess the bioequivalence between fluconazole 50mg capsules from two different manufacturers. This is a open-label, randomized, single dose, 2-treatment, 2-period crossover study in healthy Korean male and female subjects aged 19-55, to assess the bioequivalence after taking study drugs.

DETAILED DESCRIPTION:
Twenty-eight (28) healthy subjects will be enrolled into the study. Screening evaluation will occur within 28 days prior to the first dose of study medication.

Subjects will be randomized to the following treatments:

* Treatment A: Fluconazole capsule, 1 x 50 mg, Diflucan, West Ryde (REFERENCE)
* Treatment B: Fluconazole capsule, 1 x 50 mg, Diflucan, Amboise (TEST)

ELIGIBILITY:
Inclusion Criteria

* Healthy male and subjects who are between the ages of 19 and 55 years.
* Female subjects who are found not to be pregnant in physical examinations
* BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
* Subjects who are willing and able to comply with all study procedures.

Exclusion Criteria

* Evidence or history of clinically significant disease
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug test.
* History of regular alcohol consumption exceeding standard for the study
* Treatment with an investigational drug within 3 months or 5 half-lives preceding the first dose of investigational product (whichever is longer).
* Screening seated BP 140 mm Hg (systolic) or 90 mm Hg (diastolic) and over
* Screening supine 12-lead ECG demonstrating a corrected QT (QTc) interval over 450 msec or a QRS interval over 120 msec.
* Subjects with ANY of the following abnormalities in clinical laboratory tests at screening, when assessed by the study-specific laboratory and confirmed by a single repeat test:

  • Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level over 2 upper limit of normal (ULN); Total bilirubin level 2.0 mg/mL and over; subjects with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is same or under ULN.
* Pregnant female subjects, breastfeeding female subjects, male subjects, who are fertile enough and female subjects of childbearing potential for at least 28 days after the last dose of investigational product.
* Use of prescription or nonprescription drugs and dietary supplements within 10 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product.
* Use of any drugs known to significantly induce (e.g., barbiturates) or inhibit drug- metabolizing enzymes or excessive alcohol consumption within one month prior to the time of screening.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of hepatitis B surface antigen (HBsAg), hepatitis C antibody (anti-HCV), human immunodeficiency virus (HIV) antigen or antibody, and/or syphilis (RPR, Rapid Plasma Reagin test).
* Unwilling or unable to comply with the criteria in the Lifestyle Requirements section of this protocol.
* Subjects who are investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
* Other acute or chronic medical or psychiatric condition
* Subjects with known sensitivity to the drug or any of the insert ingredients or to related azole compounds.
* Subjects with hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

PRIMARY OUTCOMES:
1.Area Under Curve [AUC]last of fluconazole in Whole blood | At pre-dose (immediately prior to dosing) and 0.16, 0.33, 0.75, 1, 1.5, 2, 3, 5, 8, 12, 24, 48, 72 and 96 hours postdose.
  Area Under Curve(AUC) will be evaluated with Winnonlin analysis(Linear trapezoidal linear interpolation).
2.Maximum Plasma Concentration [Cmax] of fluconazole in Whole blood | At pre-dose (immediately prior to dosing) and 0.16, 0.33, 0.75, 1, 1.5, 2, 3, 5, 8, 12, 24, 48, 72 and 96 hours postdose.
  Plasma concentrations of fluconazole will be assayed by a validated LC- MS/MS method.

SECONDARY OUTCOMES:
1.AUCinf | At pre-dose (immediately prior to dosing) and 0.16, 0.33, 0.75, 1, 1.5, 2, 3, 5, 8, 12, 24, 48, 72 and 96 hours postdose.
  Area under the plasma concentration-time profile from time zero extrapolated to infinite time
2.AUCt/AUCinf | At pre-dose (immediately prior to dosing) and 0.16, 0.33, 0.75, 1, 1.5, 2, 3, 5, 8, 12, 24, 48, 72 and 96 hours postdose.
  AUCt: Area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration (Clast) AUCinf: Area under the plasma concentration-time profile from time zero extrapolated to infinite time
3.t½ | At pre-dose (immediately prior to dosing) and 0.16, 0.33, 0.75, 1, 1.5, 2, 3, 5, 8, 12, 24, 48, 72 and 96 hours postdose.
  Half-life time of fluconazole
4.Tmax | At pre-dose (immediately prior to dosing) and 0.16, 0.33, 0.75, 1, 1.5, 2, 3, 5, 8, 12, 24, 48, 72 and 96 hours postdose.
  Time of Max concentration of fluconazole

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Chungnam National University Hospital, Clinical Trials Center, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0561026&StudyName=AN+OPEN-LABEL%2C+RANDOMIZED%2C+SINGLE+DOSE%2C+CROSSOVER+PIVOTAL+BIOEQUIVALENCE+STUDY+OF+FLUCONAZOLE+CAPSULE+50+MG+IN+HEALTHY+ADULT+SUBJECTS